CLINICAL TRIAL: NCT00390013
Title: Vulvar Pain: Treatment Trial Using Gabapentin-placebo in a Cross-over Design, Pilot Study.
Brief Title: To Evaluate if the Medication Gabapentin Lessens Vulvar Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Colleen Stockdale (Other)
Responsible Party: Sponsor-Investigator, Colleen Stockdale, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 20060674; RR00059 (Other: University of Iowa); 200606748 (Other: University of Iowa)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Vulvar Pain Symptoms; Vulvodynia (Chronic Vulvar Pain)
Keywords: Vulvar Pain
MeSH Terms: conditions — Vulvodynia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Active Comparator): Gabapentin (Neurontin) titration and dosing for total of 8 weeks (Cross over)
  Interventions: Drug: Gabapentin
- Placebo oral capsule (Placebo Comparator): Placebo titration and dosing for total of 8 weeks (Cross over)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Gabapentin — 300 mg. capsules
  Dosage schedule for weeks 1 and 2 and weeks 12 and 13:
  1. day 1 you will take 1 capsule for the day
  2. day 2 you will take 1 capsule 2 times for that day
  3. days 3-6 you will take 1 capsule 3 times for those days
  4. days 7-9 you will take 1 capsule in am and 1 capsule at noon, 2 capsules at bedtime each day
  5. days 10-12 you will take 1 capsule in am and 2 capsules at noon and 2 capsules at bedtime each day
  6. days 13-14 you will take 2 capsules 3 times each day
  7. continue on 2 capsules 3 times each day for 6 weeks after maximum dose of 1800 mg is reached after weeks 2 and 13.
  8. at completion of study treatment you will titrate off study drug over a weeks time.
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo oral capsule — Placebo capsules
  Dosage schedule for weeks 1 and 2 and weeks 12 and 13:
  1. day 1 you will take 1 capsule for the day
  2. day 2 you will take 1 capsule 2 times for that day
  3. days 3-6 you will take 1 capsule 3 times for those days
  4. days 7-9 you will take 1 capsule in am and 1 capsule at noon, 2 capsules at bedtime each day
  5. days 10-12 you will take 1 capsule in am and 2 capsules at noon and 2 capsules at bedtime each day
  6. days 13-14 you will take 2 capsules 3 times each day
  7. continue on 2 capsules 3 times each day for 6 weeks after maximum dose of 1800 mg is reached after weeks 2 and 13.
  8. at completion of study treatment you will titrate off study drug over a weeks time.
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
The purpose of this research study is to evaluate if the medication gabapentin lessens the vulvar pain some women experience.

DETAILED DESCRIPTION:
There is not a "best" treatment plan for vulvar pain including vulvodynia (chronic vulvar pain) and vulvar vestibulitis syndrome (VVS, chronic vulvar pain localized to the vaginal opening). We propose that vulvodynia is a neuropathic pain (pain that effects the nervous system) as characterized by pain from stimuli that is not usually painful, stimuli that would not usually be painful causing significant pain, and burning pain. Gabapentin has been shown to be effective in treating chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* All women, ages 18 years and older with the diagnosis of vulvodynia or VVS (by Friedrich's criteria), who present to the University of Iowa Vulvar Vaginal Disease Clinic.

Exclusion Criteria:

* Vulvar Vaginal Disease clinic patients who are pregnant, less than 3 months postpartum, breast-feeding, non-English speaking, or have contraindication to use of gabapentin due to allergy or renal disease (serum creatinine level greater than 1.4).

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kennedy Stockdale, M.D., M.S., Principal Investigator — University of Iowa Hospital and Clinics, Department of Ob/Gyn
Locations (1):
- University of Iowa Hospital and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study has 2 phases:
  first was a placebo controlled randomized study (4 participants) second was a cross-over study (5 participants - 2 did not cross over)
Groups:
- Gabapentin First Then Placebo Crossover: Gabapentin (Neurontin) titration and dosing for total of 8 weeks (Cross over)
  Gabapentin: 300 mg. capsules
  Dosage schedule for weeks 1 and 2 and weeks 12 and 13:
  1. day 1 you will take 1 capsule for the day
  2. day 2 you will take 1 capsule 2 times for that day
  3. days 3-6 you will take 1 capsule 3 times for those days
  4. days 7-9 you will take 1 capsule in am and 1 capsule at noon, 2 capsules at bedtime each day
  5. days 10-12 you will take 1 capsule in am and 2 capsules at noon and 2 capsules at bedtime each day
  6. days 13-14 you will take 2 capsules 3 times each day
  7. continue on 2 capsules 3 times each day for 6 weeks after maximum dose of 1800 mg is reached after weeks 2 and 13.
  8. at completion of cross-over period 1 you will titrate off study drug over a weeks time.
  Placebo:
  Dosage schedule for cross-over period 2 is the same protocol as cross-over period 1 (gabapentin).
- Placebo Oral Capsule First Then Gabapentin Crossover: Placebo titration and dosing for total of 8 weeks (Cross over)
  Placebo oral capsule: Placebo capsules
  Dosage schedule for weeks 1 and 2 and weeks 12 and 13:
  1. day 1 you will take 1 capsule for the day
  2. day 2 you will take 1 capsule 2 times for that day
  3. days 3-6 you will take 1 capsule 3 times for those days
  4. days 7-9 you will take 1 capsule in am and 1 capsule at noon, 2 capsules at bedtime each day
  5. days 10-12 you will take 1 capsule in am and 2 capsules at noon and 2 capsules at bedtime each day
  6. days 13-14 you will take 2 capsules 3 times each day
  7. continue on 2 capsules 3 times each day for 6 weeks after maximum dose of 1800 mg is reached after weeks 2.
  8. at completion of study treatment (week 11) you will titrate off study drug over a weeks time.
  Gabapentin: 300 mg. capsules Dosage schedule for cross-over period 2 is the same protocol as cross-over period 1 (placebo).
- Treatment Only (Gabapentin): 1st phase (placebo controlled study) gabapentin 1800 mg max dose
- Placebo Control Arm: 1 phase Placebo
Period: Phase 1
Arm/Group | Gabapentin First Then Placebo Crossover | Placebo Oral Capsule First Then Gabapentin Crossover | Treatment Only (Gabapentin) | Placebo Control Arm
Started | 0 | 0 | 2 | 2
Completed | 0 | 0 | 2 | 1
Not Completed | 0 | 0 | 0 | 1
Not completed — tired | 0 | 0 | 0 | 1
Period: Phase 2 First Treatment
Arm/Group | Gabapentin First Then Placebo Crossover | Placebo Oral Capsule First Then Gabapentin Crossover | Treatment Only (Gabapentin) | Placebo Control Arm
Started | 3 | 2 | 0 | 0
Completed | 2 | 1 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — tired | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Phase 2 Second Treatment
Arm/Group | Gabapentin First Then Placebo Crossover | Placebo Oral Capsule First Then Gabapentin Crossover | Treatment Only (Gabapentin) | Placebo Control Arm
Started | 2 | 1 | 0 | 0
Completed | 2 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Cross Over Participants: Gabapentin (Neurontin) titration and dosing for total of 8 weeks (Cross over)
  Gabapentin: 300 mg. capsules
  Dosage schedule for weeks 1 and 2 and weeks 12 and 13:
  1. day 1 you will take 1 capsule for the day
  2. day 2 you will take 1 capsule 2 times for that day
  3. days 3-6 you will take 1 capsule 3 times for those days
  4. days 7-9 you will take 1 capsule in am and 1 capsule at noon, 2 capsules at bedtime each day
  5. days 10-12 you will take 1 capsule in am and 2 capsules at noon and 2 capsules at bedtime each day
  6. days 13-14 you will take 2 capsules 3 times each day
  7. continue on 2 capsules 3 times each day for 6 weeks after maximum dose of 1800 mg is reached after weeks 2 and 13.
  8. at completion of study treatment you will titrate off study drug over a weeks time.
  Placebo:
  Dosage schedule for cross-over period 2 is the same protocol as cross-over period 1 (Gabapentin).
- Total: Total of all reporting groups
Arm/Group | All Cross Over Participants | Gabapentin (Phase 1) | Placebo (Phase 1) | Total
Number analyzed (Participants) | 5 | 2 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 2 | 9
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 9
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 2 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 2 | 2 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Vulvar Pain
Description: change in vulvar pain following gabapentin compared to placebo - will evaluate the efficacy of gabapentin to decrease vulvar pain compared to placebo. end of 1st treatment (after 8 weeks) and end of 2nd treatment (after 19 weeks). Pain was assessed using ordinal scale (0-10): 0 = no pain, 10 = most severe pain.
Time Frame: 19 weeks
Population: study terminated early due to poor recruitment
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | -1.3 [-6 to 0] | -1.3 [-5 to 0]

ADVERSE EVENTS:
Description: participants who received the treatments were monitored
Groups:
- Gabapentin: Gabapentin (Neurontin) titration and dosing for total of 8 weeks (Cross over)
  Gabapentin: 300 mg. capsules
  Dosage schedule for weeks 1 and 2 and weeks 12 and 13:
  1. day 1 you will take 1 capsule for the day
  2. day 2 you will take 1 capsule 2 times for that day
  3. days 3-6 you will take 1 capsule 3 times for those days
  4. days 7-9 you will take 1 capsule in am and 1 capsule at noon, 2 capsules at bedtime each day
  5. days 10-12 you will take 1 capsule in am and 2 capsules at noon and 2 capsules at bedtime each day
  6. days 13-14 you will take 2 capsules 3 times each day
  7. continue on 2 capsules 3 times each day for 6 weeks after maximum dose of 1800 mg is reached after weeks 2 and 13.
  8. at completion of study treatment you will titrate off study drug over a weeks time.
- Placebo Oral Capsule: Placebo titration and dosing for total of 8 weeks (Cross over)
  Placebo oral capsule: Placebo capsules
  Dosage schedule for weeks 1 and 2 and weeks 12 and 13:
  1. day 1 you will take 1 capsule for the day
  2. day 2 you will take 1 capsule 2 times for that day
  3. days 3-6 you will take 1 capsule 3 times for those days
  4. days 7-9 you will take 1 capsule in am and 1 capsule at noon, 2 capsules at bedtime each day
  5. days 10-12 you will take 1 capsule in am and 2 capsules at noon and 2 capsules at bedtime each day
  6. days 13-14 you will take 2 capsules 3 times each day
  7. continue on 2 capsules 3 times each day for 6 weeks after maximum dose of 1800 mg is reached after weeks 2 and 13.
  8. at completion of study treatment you will titrate off study drug over a weeks time.
Arm/Group | Gabapentin | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Lack of enrollment leading to early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes